CLINICAL TRIAL: NCT04274387
Title: The Neurophysiological Effect of Mindfulness-Based Stress Reduction (MBSR) Training on Emotional Regulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201803115RINC
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Mindfulness-based Stress Reduction
Keywords: cognitive reappraisal, mindfulness, emotion regulation, emotional distress
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: one group took MBSR course the other group serve as passive control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR group (Experimental): participants who receiving 8-week MBSR between the pretest and posttest
  Interventions: Behavioral: Mindfulness-based Stress Reduction(MBSR)
- passive control group (No Intervention): participants who not undergoing any interventions for 8 weeks between the pretest and posttest

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction(MBSR) — A structural program focusing on the practice about attending to the current moment with non-judgmental attitude
  Arms: MBSR group

SUMMARY:
Background Emotional distress is known to render vicious effects both mentally and physiologically to human beings. Emotional regulation is therefore an important capability to dilute the poisonous effect of emotional distress. The cognitive reappraisal and mindfulness thinking are two major strategies that have been empirically tested and supported to be effective emotional regulation approaches. Oftentimes, entry-level practitioners of mindfulness get confused easily between the cognitive reappraisal and mindfulness approach to emotional regulation in that they look similar in some of their practice forms. However, they are quite different from each other in terms of their fundamental concept. Although there are already many studies contribute to the mechanisms underlying these two approaches independently, very few studies have been proposed to directly investigate the fundamental differences of the underlying neural mechanisms between the two approaches. The current proposal therefore aims to compare the underlying neural mechanisms between the cognitive reappraisal and the mindfulness approaches within the context of emotional processing.

Objectives We propose herein a 2-year research project to address the following two hypotheses: (1) we hypothesize that the differences in terms of neural activation patterns between the mindfulness and cognitive reappraisal responses toward positive or negative stimuli in the emotion regulation task (ERT) will appear only after certain amount of MBSR training and (2) we hypothesize that the 10-week Mindfulness-based Stress Reduction (MBSR) training will be accompanied by the increased resting-state functional connectivity between the salience network (involved in the process of meta-awareness) and both the dorsal attention network (i.e., attention to the outside world) and the default mode network (i.e., attention to the internal state).

Methods For the current proposal, we will use a pre-post-test plus longitudinal follow-up design research design. Based on the power analysis, we expect to recruit 45 adults (convenient sampling). We will collect neuropsychological, EEG and fMRI data from each participants at three time points with one time point before the MBSR training course (pre-test), one time point immediately after completing the MBSR training course (post-test) and one time point 8 months after completing the MBSR training course (8-month follow-up). For the neuropsychological measures, we will use the MAAS for evaluating trait mindfulness, DERS for evaluating emotional regulation and dysregulationand IRI for evaluating cognitive and emotional empathy level. For the fMRI measures, we will analyze the functional activation patterns between the cognitive reappraisal and the mindfulness process of emotion regulation. Furthermore, we will analyze the functional connectivity based on the resting-state fMRI data to investigate the change of pre- and post-MBSR training. For EEG measures, we will further analyze the different time-frequency patterns between these two types of emotional regulation.

Anticipated results We expect that the results will help unravel the functional changes of neuronal circuits associated with the transition from habitual cognitive reappraisal strategy to a mindfulness strategy, after an intensive mindfulness-based training. We hope that the overall outcomes from the current proposal will help enrich our knowledge that will enhances the translation of applying cognitive reappraisal and mindfulness based approaches in clinical psychiatry.

Keywords: cognitive reappraisal, mindfulness, emotion regulation, emotional distress

ELIGIBILITY:
Inclusion Criteria: (1) aged 20~60 years and over; (2) no a-prior experience of any form of mindfulness/meditation training (3) being able to understand and speak Taiwanese or Mandarin; (4) no participation in any drug studies during this project period.

Exclusion Criteria: (1) aged over 60 or under 20; (2) have been trained with any form of mindfulness/meditation; (3) not speaking Taiwanese or Mandarin; (4) an inability to understand the survey questions due to apparent cognitive difficulties, serious deficits in vision or hearing; and (5) medical history of psychiatric disorders and neurological diseases (measured with BSRS-30) ;(6) have metal implants placed in the body;(7) have contraindications for undergoing an MRI scan such as having a heart pacemaker or an artificial heart valve, history of having a metal sliver in the eye or an aneurysm clip in their brain, having implanted surgical clips, having claustrophobia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-14 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
psychological trait change | within a month
  measured by related questionnaire
subjective rating in valence/ arousal of emotional pictures | within a month
  measured subjects' behavior emotion response in valence and arousal toward IAPS pictures
EEG-derived index, Late Positive Potential (LPP) | within a month
  measured subjects' neural emotion process toward IAPS pictures

CONTACTS AND LOCATIONS:
Locations (1):
- School of Occupational Therapy, College of Medicine National Taiwan University, Taipei, Taiwan